CLINICAL TRIAL: NCT00225927
Title: A Prospective, Randomized, Controlled Trial of Radioguided Seed Localization Versus Standard Needle Localization of Nonpalpable Breast Cancers
Brief Title: Trial Comparing Radioactive Seed Localization to Standard Procedure for Non-palpable Breast Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Dr. Peter J. Lovrics, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2005-09-16; First posted 2005-09-26 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Breast Cancer Invasive Nos; Stage 0 Breast Carcinoma
Keywords: invasive breast cancer; in situ breast cancer; radioguided seed localization; nonpalpable tumour; needle localization; margin status
MeSH Terms: conditions — Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: radioguided seed localization for nonpalpable breast cancers — radio-labelled (I-125) titanium seed inserted via needle into nonpalpable breast lesion and gamma probe used to guide surgery

SUMMARY:
The purpose of this study is to determine whether a new surgical technique (radioguided seed localization) for localizing nonpalpable breast tumours is better than the standard technique (needle localization).

DETAILED DESCRIPTION:
Most breast cancers are removed by partial mastectomy/lumpectomy. The most important factor in ensuring that the cancer does not return in the breast is to ensure that it is completely removed during surgery. Complete removal is dependent on having a rim of normal tissue (clear margin) surrounding the cancer. If the margin is positive, or the cancer recurs, more surgery or mastectomy is required. Approximately one third of breast cancers are detected by mammograms or ultrasounds and cannot be felt by patients or physicians. Accordingly, a localization technique is required to help the surgeon to find and remove the cancer. The current technique (needle localization) has a higher chance of having cancer cells at the margin. This is a study about a surgical technique. The objective of this comparison study is to determine whether a new technique (radioguided seed localization) is a better way to remove nonpalpable breast cancers. The main objective of this study is to determine if the new technique generates fewer positive margins compared to the standard technique. An improved technique would benefit thousands of women every year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive or in situ breast carcinoma
* Nonpalpable breast tumour
* Candidate for breast conserving surgery (BCS) based on clinical and radiologic evaluation

Exclusion Criteria:

* Histological confirmation more than 3 months from enrollment
* Pregnancy or lactation
* Contraindication to BCS or patient requests mastectomy
* Age less than 18 years
* Male patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2004-06; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Compare the number of positive margins following excision of the nonpalpable breast tumours for the two different surgical techniques | immediate post-operative pathology results

SECONDARY OUTCOMES:
Compare procedure times, complications and volume of tissue excised for both techniques | intra-operative

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Lovrics, MD, Principal Investigator — McMaster University; Mary Townsend, Study Chair — Administrator for Research Programs, McMaster University
Locations (3):
- Canada (3):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Reedijk M, Hodgson N, Gohla G, Boylan C, Goldsmith CH, Foster G, Cornacchi SD, McCready D, Lovrics PJ. A prospective study of tumor and technical factors associated with positive margins in breast-conservation therapy for nonpalpable malignancy. Am J Surg. 2012 Sep;204(3):263-8. doi: 10.1016/j.amjsurg.2012.03.007. Epub 2012 Jul 12. PMID 22794705
- [Derived] Lovrics PJ, Goldsmith CH, Hodgson N, McCready D, Gohla G, Boylan C, Cornacchi S, Reedijk M. A multicentered, randomized, controlled trial comparing radioguided seed localization to standard wire localization for nonpalpable, invasive and in situ breast carcinomas. Ann Surg Oncol. 2011 Nov;18(12):3407-14. doi: 10.1245/s10434-011-1699-y. Epub 2011 Apr 30. PMID 21533657